CLINICAL TRIAL: NCT02487576
Title: Interplay of Peripheral Circadian Clocks With Energy Balance and Body Weight Regulation
Brief Title: The CLOCK Study - A Human Dietary Intervention Study on Peripheral Circadian Clocks and Energy Metabolism
Acronym: CLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Charite University, Berlin, Germany (Other); Heidelberg University (Other); Max-Planck Institute of Molecular Cell Biology and Genetics (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Prof. Dr. med Andreas F.H. Pfeiffer, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DFG grant KFO218 PF164/16-1; DDG021023 (Other Grant/Funding Number: Deutsche Diabetes Gesellschaft)
Record Dates: First submitted 2015-05-28; First posted 2015-07-01 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Response to Dietary Modification
MeSH Terms: interventions — salmon gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate-rich_Fat-rich (HC_HF) (Other): Isocaloric carbohydrate-rich meals in the morning (06.00 am - 01.30 pm) and isocaloric fat-rich meals in the evening (04.30 pm - 10.00 pm) for 4 weeks
- Fat-rich_Carbohydrate-rich (HF_HC) (Other): Isocaloric fat-rich meals in the morning (06.00 am - 01.30 pm) and isocaloric carbohydrate-rich meals in the evening (04.30 pm - 10.00 pm) for 4 weeks
  Interventions: Other: Carbohydrate-rich (HC); Other: Fat-rich (HF)

INTERVENTIONS:
Other: Carbohydrate-rich (HC) — 65% Carbohydrate; 20% Fat; 15% Protein
  Arms: Fat-rich_Carbohydrate-rich (HF_HC)
Other: Fat-rich (HF) — 35% Carbohydrate; 50% Fat; 15% Protein
  Arms: Fat-rich_Carbohydrate-rich (HF_HC)

SUMMARY:
This human dietary intervention study with a cross-over design aims to investigate the effect of two different diurnal patterns of meal composition on peripheral circadian clocks and energy metabolism in healthy men.

DETAILED DESCRIPTION:
In this cross-over study, healthy male participants are randomly allocated to one of two study groups: In study group (A) participants consume isocaloric carbohydrate-rich meals (65% Carbohydrates; 20% Fat; 15% Protein) in the morning and fat-rich meals (35% Carbohydrate; 50% Fat; 15% Protein) in the evening for four weeks. After a washout-phase participants consume isocaloric fat-rich meals in the morning and carbohydrate-rich meals in the evening for another four weeks. Study group (B) receives the same interventions in the reversed order.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 22 kg/m² and 34,9 kg/m²
* Normal glucose tolerance determined in a 75g-oral glucose tolerance test
* Impaired fasting glucose determined in a 75g-oral glucose tolerance test
* Impaired glucose tolerance determined in a 75g-oral glucose tolerance test

Exclusion Criteria:

* Shift workers or history of shift work
* Men suffering from diseases or conditions that might influence the outcome of the study. Of special interest are diseases that influence body weight regulation (enteropathy, malabsorption, hepatopathy, renal disease, endocrine disorders, diabetes mellitus, eating disorders, heart disease etc.). Also men suffering from coagulopathy, apoplexy and myocardial infarction are excluded from the study.
* Men suffering from psychiatric disease
* Planned changes in physical activity during the study
* Participation in other clinical studies within the last three months
* Weight changes > 2 kg within 2 months prior to screening day
* Men unable to give an informed consent
* Men unable to engage in the dietary interventions
* Men following a special diet

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Dietary-induced changes of glucose and lipid metabolism | week 4
Effect of different diurnal patterns of meal composition on peripheral circadian clocks in blood cells and subcutaneous adipose tissue | week 4

SECONDARY OUTCOMES:
Dietary-induced changes of satiety and hunger scores | week 4
  Measured via visual analogue scales
Effect of different diurnal patterns of meal composition on Lipopolysaccharide-induced cytokine expression | week 4
Dietary-induced changes of the human adipose tissue lipidome | week 4
Integrative analysis of dietary-induced changes of the human adipose tissue transcriptome | week 4
  Microarray Analysis of adipose tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof. Dr., Study Director — German Institute of Human Nutrition
Locations (1):
- German Institute of Human Nutrition, Potsdam, Germany

REFERENCES:
- [Background] Kessler K, Hornemann S, Petzke KJ, Kemper M, Kramer A, Pfeiffer AF, Pivovarova O, Rudovich N. The effect of diurnal distribution of carbohydrates and fat on glycaemic control in humans: a randomized controlled trial. Sci Rep. 2017 Mar 8;7:44170. doi: 10.1038/srep44170. PMID 28272464
- [Background] Kessler K, Hornemann S, Petzke KJ, Kemper M, Markova M, Rudovich N, Grune T, Kramer A, Pfeiffer AFH, Pivovarova-Ramich O. Diurnal distribution of carbohydrates and fat affects substrate oxidation and adipokine secretion in humans. Am J Clin Nutr. 2018 Dec 1;108(6):1209-1219. doi: 10.1093/ajcn/nqy224. PMID 30541098
- [Background] Kessler K, Gerl MJ, Hornemann S, Damm M, Klose C, Petzke KJ, Kemper M, Weber D, Rudovich N, Grune T, Simons K, Kramer A, Pfeiffer AFH, Pivovarova-Ramich O. Shotgun Lipidomics Discovered Diurnal Regulation of Lipid Metabolism Linked to Insulin Sensitivity in Nondiabetic Men. J Clin Endocrinol Metab. 2020 May 1;105(5):dgz176. doi: 10.1210/clinem/dgz176. PMID 31680138
- [Background] Kessler K, Hornemann S, Rudovich N, Weber D, Grune T, Kramer A, Pfeiffer AFH, Pivovarova-Ramich O. Saliva Samples as A Tool to Study the Effect of Meal Timing on Metabolic And Inflammatory Biomarkers. Nutrients. 2020 Jan 28;12(2):340. doi: 10.3390/nu12020340. PMID 32013045